CLINICAL TRIAL: NCT01591122
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Study of Abiraterone Acetate (JNJ-212082) Plus Prednisone in Asymptomatic or Mildly Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of Abiraterone Acetate Plus Prednisone in Patients With Chemo-naive Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100011; ABI-PRO-3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Metastatic Castration Resistant Prostate Cancer; Abiraterone acetate; Prednisone; Zytiga
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Abiraterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abiraterone acetate and prednisone (Experimental)
  Interventions: Drug: Abiraterone acetate and prednisone
- Placebo and prednisone (Active Comparator)
  Interventions: Drug: Placebo and prednisone

INTERVENTIONS:
Drug: Placebo and prednisone — Placebo: Form=tablet, route=oral. Four tablets daily on an empty stomach. Prednisone: Type=exact number, unit=mg, number=5, form=tablet, route=oral, twice daily.
  Arms: Placebo and prednisone
Drug: Abiraterone acetate and prednisone — Abiraterone acetate: Type=exact number, unit=mg, number=250, form=tablet, route=oral. Four tablets daily on an empty stomach Prednisone: Type=exact number, unit=mg, number=5, form=tablet, route=oral, twice daily
  Arms: Abiraterone acetate and prednisone

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of abiraterone acetate when co-administered with prednisone in patients with chemo-naive metastatic castration resistant prostate Cancer (mCRPC).

DETAILED DESCRIPTION:
This is a multinational, multicenter, randomized (the study drug is assigned by chance), double-blind (neither physician nor patient knows the treatment that the patient receives), placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) study. All patients will be randomly assigned in a 1:1 ratio between the abiraterone acetate group (abiraterone acetate and prednisone) and the placebo group (placebo and prednisone). The study will consist of a screening phase (within 28 days prior randomization on Cycle 1, Day 1), a treatment phase (28-day cycles until disease progression), and a follow-up phase (all patients will be contacted for every 3 months up to Month 60, focusing primarily on survival status). Patients will receive either abiraterone acetate 1,000 mg daily and prednisone 5 mg twice daily or placebo and prednisone 5 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of adenocarcinoma of the prostate with evidence of metastatic disease
* Prostate cancer progression documented by PSA progression or radiographic progression
* Asymptomatic or mildly symptomatic from prostate cancer
* Surgically or medically castrated, with testosterone levels of <50 ng/dL
* Previous anti-androgen therapy and progression after withdrawal
* ECOG performance status score of 0 or 1
* If opiate analgesics for cancer-related pain, treatment must not be administered within 4 weeks of Cycle 1 Day 1
* If radiation therapy for treatment of the primary tumor is given, treatment must not be administered within 6 weeks of Cycle 1 Day 1
* If previously treated with ketoconazole for prostate cancer, duration of treatment must not be greater than 7 days
* Life expectancy of at least 6 months

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone (corticosteroid) use contraindicated
* Any chronic medical condition requiring a higher dose of corticosteroid than 5 mg prednisone twice daily
* Pathological finding consistent with small cell carcinoma of the prostate
* Liver or visceral organ metastasis, brain metastasis, and other malignancy, except non-melanoma skin cancer, with a 30% probability of recurrence within 24 months
* Prior cytotoxic chemotherapy or biologic therapy for the treatment of metastatic castration-resistant prostate cancer (mCRPC)
* Radiation or radionuclide therapy for treatment of mCRPC
* Uncontrolled hypertension, patients with a history of hypertension are allowed provided blood pressure is controlled by anti hypertensive treatment
* History of pituitary or adrenal dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Time to prostate specific antigen (PSA) progression (TTPP) | 14 months
  Measured from the time interval from the date of randomization to the date of the PSA progression based on prostate cancer clinical trials working group 2 (PCWG2) criteria

SECONDARY OUTCOMES:
Overall survival | 5 years
  The percentage of people in a study or treatment group who are alive from date of randomization to date of death
Time to initiation of cytotoxic chemotherapy | 5 years
  Date of randomization to date of initiation of chemotherapy
Prostate specific antigen (PSA) response rate | 14 months
  Proportion of patients achieving a PSA decline 50% according to prostate cancer clinical trials working group 2 (PCWG2) criteria
Objective response rate | 14 months
  Measurable disease based on modified response evaluation criteria in solid tumors (RECIST) criteria and baseline lymph node size must be 2.0 cm to be considered target or evaluable lesion for RECIST criteria
Quality of life (QoL) total score and each subscale score | 14 months
  Assessed by functional assessment of cancer therapy-prostate (FACT-P)
Time to pain progression | 14 months
  Assessed by the Brief Pain Inventory Short Form (BPI-SF) and analgesic score
Time to Eastern Cooperative Oncology Group (ECOG) performance status score determination | 14 months
  ECOG performance status score 0 (Fully active, able to carry on all pre-disease performance without restriction) versus 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work on a light or sedentary nature, eg, light housework, office work)
Collection of safety data including adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (22):
- China (10):
  - Beijing
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Jinan
  - Nanjing
  - Shanghai
  - Tianjin
  - Wuhan
- Kuala Lumpur, Malaysia
- Russia (10):
  - Arkhangelsk
  - Moscow
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Sochi
  - Stavropol
  - Ufa
  - Yekaterinburg
  - Yoshkar-Ola
- Bangkok, Thailand

REFERENCES:
- See also: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Abiraterone Acetate (JNJ-212082) Plus Prednisone in Asymptomatic or Mildly Symptomatic Patients with Metastatic Castration-Resistant Prostate Cancer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR100011&attachmentIdentifier=1f6dad2c-ce67-418a-b152-d8a1f9847a97&fileName=CR100011_CSR_Synopsis.pdf&versionIdentifier=